CLINICAL TRIAL: NCT02826993
Title: Can Colon Capsule Endoscopy Substitute CT Colonography in the Large Bowel Examination of Persons Whose Colonoscopy Was Incomplete?
Brief Title: Patients With Incomplete Colonoscopy a Comparison of Colon Capsule Endoscopy and CT Colonography
Acronym: CfC100
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Morten Kobaek-Larsen, Project Coordinator, Odense University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OdenseUH_MKL1
Record Dates: First submitted 2016-05-20; First posted 2016-07-11 (Estimated); Last update posted 2021-09-10 (Actual); Status verified 2018-08

CONDITIONS: Incomplete Colonoscopy; CT Colonography; Camera Capsule Endoscopy
Keywords: PillCAM2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CCE in incomplete Colonoscopies (Experimental): Patients in which colonoscopy is not possible are invited for CT colonography and those patients are examined by Camera Capsule Endoscopy the day before the CT colonography and the two different examinations are compared.
  Interventions: Device: CCE in incomplete Colonoscopies

INTERVENTIONS:
Device: CCE in incomplete Colonoscopies — When the initial colonoscopy has failed, participants are invited to ingest a CCE on the day prior to their subsequent CT colonography. Thus, the CCE and CT will be compared within subjects for their ability to identify and estimate sizes of polyps
  Other Names: PillCams2

SUMMARY:
A total of 8000 colonoscopies are performed on a yearly basis on the Funen Island. Between 5% and 10% of those are incomplete due to excessive pain, fixed colon loops, and other reasons. The current standard procedure is to refer the patient to the department of radiology for a CT-colonography. In some instances the radiology department can offer the investigation the next day, and thus in the same colon preparation. At other times they cannot, and the patient has to go through an second colon preparation for the colonography.

A CCE procedure could be provided to the participants immediately after the failed colonoscopy and the investigation can be completed the next morning in the same bowel preparation without a visit to the radiology department.

DETAILED DESCRIPTION:
Optical colonoscopy is the standard method for evaluating the colon. This technique allows evaluation of the entire colon in most patients. Full colonoscopy including examination of the cecum is associated with an increased detection rate of advanced neoplasia, as 33-50% of advanced neoplasia is located in the proximal colon. After an incomplete optical colonoscopy, participants are required to undergo another test in order to exclude clinically relevant lesions to reduce the risk of proximal cancer which has been shown to increase by twofold when colonoscopy was incomplete.

Endoscopic and radiological options to complete the colon assessment have been available in the last decades. Multiple alternative endoscopic techniques-such as colonoscopy with thinner colonoscopes, gastroscopes and device-assisted enteroscopes have been described. However, none of them has been clearly standardized.

CT colonography (CTC), is a relatively new imaging technique that was first described in 1994. In large randomized trials on symptomatic patients, CTC has been shown to be as equally effective as colonoscopy - for the detection of large colorectal polyps and already developed colorectal cancer.

Colon Capsule Endoscopy (CCE) is a promising new technology that may have the potential to complement existing diagnostic methods to screen people for colorectal cancer. Delivered correctly, it may reduce costs, increase utilization of medical services, reduce risks for patients and overall improve screening rates among the population.

A total of 8000 colonoscopies are performed on a yearly basis on the Funen Island and about 10% of those are incomplete due to excessive pain, fixed colon loops, and others causes. The current standard procedure is to refer the participant to the Department of Radiology for a CT-colonography.

ELIGIBILITY:
Inclusion Criteria:

* Incomplete colonoscopy

Exclusion Criteria:

* Previous gastrointestinal surgery except for appendectomy
* Known inflammatory bowel disease including Crohn's disease and ulcerative colitis
* An ostomy
* Diabetes
* Symptoms on bowel obstruction
* Pacemakers
* Kidney diseases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-06; Primary Completion 2019-04-01 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of CCE compared to CTC | Up to 14 days for conducting both procedures
  The sensitivity and specificity of CCE will be measured in terms of n of polyps detected by CCE compared to n of polyps detected by CTC

SECONDARY OUTCOMES:
Size estimation | Up to 14 days for conducting both procedures
  Each polyp is estimated in terms of size through the use of both technologies
Polyp miss rate | Up to 30 days for conducting all three procedures
  The rate of polyps missed by CCE and CTC respectively compared to a colonoscopy that will be performed in full sedation for participants in whom discrepancy is found between the two modalities (CCE and CTC)

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Baatrup, Professor, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Svendborg Sygehus, Svendborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Deding U, Herp J, Havshoei AL, Kobaek-Larsen M, Buijs MM, Nadimi ES, Baatrup G. Colon capsule endoscopy versus CT colonography after incomplete colonoscopy. Application of artificial intelligence algorithms to identify complete colonic investigations. United European Gastroenterol J. 2020 Aug;8(7):782-789. doi: 10.1177/2050640620937593. PMID 32731841